CLINICAL TRIAL: NCT06045611
Title: The Effect of Oral Ingestion of Animal and Plant-based Proteins on the Somatotropic Axis
Brief Title: The Effect of Oral Intake of Animal and Plant Proteins on the Metabolism in Healthy Women
Acronym: PAN-Promet
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Dnr 2023-03852-01
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Protein; Plant-based protein; Metabolism; Somatotrophic Axis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Isolated Pea Protein/Isolated Whey Protein/Isolated Faba Bean Protein/Placebo (Experimental): * Study day 1: 0.6g isolated pea protein/kg/body weight + 400 ml water
  * Study day 2: 0.6g isolated whey protein/kg/body weight + 400 ml water
  * Study day 3: 0.6g isolated faba bean protein/kg/body weight + 400 ml water
  * Study day 4: 400 ml water
  The fat and energy content of the drinks will be adapted using a plant based oil
  Interventions: Dietary Supplement: Isolated Pea Protein; Dietary Supplement: Isolated Whey Protein; Dietary Supplement: Isolated Faba Bean Protein; Dietary Supplement: Placebo
- Isolated Whey Protein/Placebo/Isolated Pea Protein/Isolated Faba Bean Protein (Experimental): * Study day 1: 0.6g isolated whey protein/kg/body weight + 400 ml water
  * Study day 2: 400 ml water
  * Study day 3: 0.6g isolated pea protein/kg/body weight + 400 ml water
  * Study day 4: 0.6g isolated faba bean protein/kg/body weight + 400 ml water
  The fat and energy content of the drinks will be adapted using a plant based oil
  Interventions: Dietary Supplement: Isolated Pea Protein; Dietary Supplement: Isolated Whey Protein; Dietary Supplement: Isolated Faba Bean Protein; Dietary Supplement: Placebo
- Isolated Faba Bean Protein/Isolated Pea Protein/Placebo/Isolated Whey Protein (Experimental): * Study day 1: 0.6g isolated faba bean protein/kg/body weight + 400 ml water
  * Study day 2: 0.6g isolated pea protein/kg/body weight + 400 ml water
  * Study day 3: 400 ml water
  * Study day 4: 0.6g isolated whey protein/kg/body weight + 400 ml water
  The fat and energy content of the drinks will be adapted using a plant based oil
  Interventions: Dietary Supplement: Isolated Pea Protein; Dietary Supplement: Isolated Whey Protein; Dietary Supplement: Isolated Faba Bean Protein; Dietary Supplement: Placebo
- Placebo/Isolated Faba Bean Protein/Isolated Whey Protein/Isolated Pea Protein (Experimental): * Study day 1: 400 ml water
  * Study day 2: 0.6g isolated faba bean protein/kg/body weight + 400 ml water
  * Study day 3: 0.6g isolated whey protein/kg/body weight + 400 ml water
  * Study day 4: 0.6g isolated pea protein/kg/body weight + 400 ml water
  The fat and energy content of the drinks will be adapted using a plant based oil
  Interventions: Dietary Supplement: Isolated Pea Protein; Dietary Supplement: Isolated Whey Protein; Dietary Supplement: Isolated Faba Bean Protein; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Isolated Pea Protein — Participants will consume the protein supplement dissolved in water in an opaque mug wearing a nose clip.
Dietary Supplement: Isolated Whey Protein — Participants will consume the protein supplement dissolved in water in an opaque mug wearing a nose clip.
Dietary Supplement: Isolated Faba Bean Protein — Participants will consume the protein supplement dissolved in water in an opaque mug wearing a nose clip.
Dietary Supplement: Placebo — Participants will consume the placebo in an opaque mug wearing a nose clip.

SUMMARY:
The goal of this interventional study is to learn about the effects of different proteins (from animals or plants) on the metabolism in healthy, normal weight women between 18-45 year who are not on hormonal birth-control.

The main questions the study aims to answer are:

1. How do different proteins affect biological markers of the metabolism and which protein has the strongest effect?
2. How are the different proteins digested and taken up from our body?

Participants will drink four different shakes on four different study days in a random order. Three of them contain each a different protein and one does not contain protein. Right before drinking the shake and on 11 timepoints after drinking the shake blood samples will be drawn.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Age: 18-45 years
* Body mass index: 18.5 < 25 kg/m2
* Signed informed consent

Exclusion Criteria:

* Use of hormonal contraceptives
* Pregnancy or breastfeeding
* Diabetes mellitus or any other metabolic disease that might affect the results of this study
* Gastric surgery that affects digestion and uptake of protein
* Any clinically significant present or past disease/condition and medication which in the investigator's opinion could interfere with the results of the trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Release of Growth Hormone | 0-3 hours after consumption of test drink (on all 4 study days)
  The primary outcome is defined as the postprandial release of growth hormone during three hours after oral ingestion of plant-protein test drinks vs. an animal-protein test drink measured as incremental area under the curve. Growth hormone will be measured in blood samples.

SECONDARY OUTCOMES:
Release of Hormones Related to the Somatotrophic Axis | 0-3 hours after consumption of test drink (on all 4 study days)
  We will measure different hormones related to the somatotrophin axis in collected blood samples and investigate if there are differences between different protein-sources.
Kinetics of Amino Acid Uptake | 0-3 hours after consumption of test drink (on all 4 study days)
  We will measure amino acids in collected blood samples to investigate dynamics and kinetics of protein digestion/uptake of different protein sources.

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Undecided